CLINICAL TRIAL: NCT00374296
Title: A Phase II Study of MGCD0103 (MG-0103) in Patients With Acute Myelogenous Leukemia/High Risk MDS Who Are Elderly and Have Previously Untreated Disease or Who Are Adult and Have Relapsed/Refractory Disease
Brief Title: MGCD0103 in Elderly Patients With Previously Untreated AML/High Risk MDS or Adults With Relapsed/Refractory Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Clinical Development Program for MGCD0103 is being re-evaluated
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-007
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Myelogenous Leukemia, Acute; Myelodysplastic Syndromes
Keywords: Leukemia; MDS; Phase II; Acute Myelogenous Leukemia (AML); High Risk Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Elderly (≥65 years) untreated arm
- 2 (Experimental): Relapsed/Refractory Arm
  Interventions: Drug: MGCD0103

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 administered orally three-times per week
  Arms: 2

SUMMARY:
In this study, MGCD0103, a new anticancer drug under investigation, is given three times per week to elderly patients with previously untreated acute myelogenous leukemia/high risk myelodysplastic syndrome or adults with relapsed/refractory disease.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of AML or high risk MDS.
* Elderly cohort (70 years of age or more): no prior chemotherapy treatment for AML/high risk MDS and not currently candidates for intensive chemotherapy.
* Relapsed/refractory cohort (18 years of age or more): relapsed or refractory to prior treatment.
* ECOG performance status of 0 or 1.
* Total bilirubin < 1.5 x upper limit of normal (ULN).
* AST/SGOT and ALT/SGPT < 2.5 x ULN.
* Serum creatinine < 1.5 x ULN.
* Patients must read, understand, and sign a written informed consent form (ICF).
* Women of childbearing potential and male patients' female partners must use an acceptable method of contraception while on study, and for 3 months after study drug treatment.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with uncontrolled, intercurrent illness, active or uncontrolled infections, or a fever > 38.5C (not due to tumor fever) on the day of scheduled dosing.
* Patients with serious illnesses or medical conditions, including laboratory results, which, in the investigator's opinion, would interfere with a patient's participation, or with the interpretation of the results.
* Patients treated with an investigational drug within 30 days prior to study initiation.
* Known hypersensitivity to HDAC inhibitors or to any of the components of MG-0103.
* Known HIV or active hepatitis B or C.
* Any condition that may affect the patient's ability to sign the ICF and undergo study procedures.
* Any conditions that will put the patient at undue risk or discomfort as a result of adherence to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year (anticipated
Response rate | 1 year (anticipated)

SECONDARY OUTCOMES:
Progression-free survival | 1 year (anticipated)
Duration of objective response | 1 year (anticipated)
Pharmacokinetics | 1 year (anticipated)
Pharmacodynamics | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (13):
- United States (6):
  - Veterans Affairs Medical Center, Kansas City, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center - James Cancer Hospital, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Canada (7):
  - Hamilton Health Sciences - McMaster Hospital, Hamilton, Ontario
  - UHN - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Sir Mortimer Davis-Jewish General Hospital, Montreal, Quebec
  - Universite de Sherbrooke, Service d'hematologie, Sherbrooke, Quebec